CLINICAL TRIAL: NCT07178509
Title: Myocardial Perfusion in Spontaneous Coronary Artery Dissection Using Stress Contrast Echocardiography
Brief Title: A Study of SCAD Using Stress Contrast Echocardiography
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Marysia Tweet, Principal Investigator, Mayo Clinic
Other Study IDs: 24-002318; 1K23HL155506 (NIH)
Record Dates: First submitted 2025-09-02; First posted 2025-09-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Spontaneous Coronary Artery Dissection
MeSH Terms: conditions — Coronary Artery Dissection, Spontaneous | interventions — Contrast Media

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spontaneous coronary artery dissection (SCAD): Subject has a history of spontaneous coronary artery dissection (SCAD)
  Interventions: Procedure: Stress Echocardiography with Contrast
- Healthy Subjects: Subjects are healthy with no significant medical history
  Interventions: Procedure: Stress Echocardiography with Contrast

INTERVENTIONS:
Procedure: Stress Echocardiography with Contrast — Stress Echocardiography with Contrast will be used to assess heart function and blood flow response to stressors.

SUMMARY:
This study aims to fill knowledge gaps regarding microvascular perfusion and pressor response to stress among patients with history of spontaneous coronary artery dissection (SCAD) using stress contrast echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Adult >18 years old
* Patient has a history of spontaneous coronary artery dissection (SCAD) OR patient is healthy with no significant medical history

Exclusion Criteria:

* Unable to give consent
* Allergic or have a history of adverse reaction to dobutamine, the Definity® ultrasound enhancing agent, or atropine.
* Has a known or suspected hypersensitivity to perflutren and therefore cannot be given Definity®.
* Pregnant.
* Unable to interrupt breastfeeding.
* Within 3 months of a heart attack.
* Severe aortic stenosis.
* Severe, uncontrolled hypertension (>200/110 mmHg at baseline).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the clinic and community.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Change in Microvascular Function | Baseline, immediately after the Stress Echocardiography
  Microvascular Function will be determined by Microvascular Blood Flow (Liters/Minute). Microvascular Blood Flow will be measured by a stress echocardiogram with contrast. A higher Microvascular Blood Flow indicated better blood flow circulation.
Change in Blood Pressure | Baseline, immediately after the Stress Echocardiography
  Change is blood pressure will be measured by a stress echocardiogram with contrast (mmHg).
Change in Heart Rate | Baseline, immediately after the Stress Echocardiography
  Change in heart rate will be measured by a stress echocardiogram with contrast (beats per minute).

CONTACTS AND LOCATIONS:
Overall Officials: Marysia Tweet, M.D., M.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No